CLINICAL TRIAL: NCT04374448
Title: The Utility of Indocyanine Green Fluorescence in Endoscopic Sinonasal and Skull Base Surgery - A Prospective Case-Series and Feasibility Study
Brief Title: Utility of Indocyanine Green Fluorescence in Endoscopic Sinonasal and Skull Base Surgery
Acronym: NIRFICG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Paul's Sinus Centre (Other)
Responsible Party: Principal Investigator, Dr. Andrew Thamboo, MD, Assistant Clinical Professor, St. Paul's Sinus Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NIRF ICG Protocol
Record Dates: First submitted 2020-04-28; First posted 2020-05-05 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Chronic Sinusitis; Tumor of Nasal Sinus; Posterior Epistaxis; Skull Base Neoplasms
Keywords: Indocyanine Green; Endoscopic Sinus Surgery; Skullbase Surgery; Sinonasal tumors
MeSH Terms: conditions — Paranasal Sinus Neoplasms; Skull Base Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective Case-Series and Feasibility Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sinus Tumor Resection (Other): Those who are undergoing endoscopic sinonasal surgery for benign and malignant tumor removal.
  Interventions: Procedure: Sinonasal Benign or Malignant Tumor Resection
- Skull Base Surgery (Other): Those who are receiving Endoscopic Skull Base Surgery (ESBS) for minimally-invasive access for removal of skull base tumors, most commonly for ones of pituitary origin.
  Interventions: Procedure: Skull Base Surgery (Assessment of Nasoseptal Flap)
- Endoscopic Sinus Surgery (Other): Individuals with chronic rhinosinusitis (CRS) with or without polyposis that are to have endoscopic sinus surgery, a minimally invasive procedure to open the sinuses.
  Interventions: Procedure: Endoscopic Sinus Surgery
- Epistaxis Management (Other): Those who have severe nose bleeds and requires going into the operating room for management.
  Interventions: Procedure: Posterior Epistaxis Management (SPA Ligation)

INTERVENTIONS:
Procedure: Sinonasal Benign or Malignant Tumor Resection — During sinus tumor resection, margins will initially be estimated with the naked eye. Then the dye, Indocyanine Green (ICG), will be injected through the intravenous line to identify tumor margins and be compared to estimated margins.
  Arms: Sinus Tumor Resection
Procedure: Skull Base Surgery (Assessment of Nasoseptal Flap) — In this surgery, a piece of individuals septum will be used for the reconstruction. The amount of time for the flap to fluoresce Indocyanine Green (ICG) will be measured. It will be ensured that the it is still lighting up at the end of the surgery, indicating it is still receiving a good supply and ensures longevity of the flap.
  Arms: Skull Base Surgery
Procedure: Endoscopic Sinus Surgery — During the surgery, the timing of Indocyanine Green (ICG) administration to fluorescence of anterior and posterior ethmoidal artery and of the internal carotid artery will be measured.
  Arms: Endoscopic Sinus Surgery
Procedure: Posterior Epistaxis Management (SPA Ligation) — During surgery timing of Indocyanin Green (ICG) administration to fluorescence of the sphenopalatine artery will be measured.
  Arms: Epistaxis Management

SUMMARY:
The endoscope is a device placed into the nasal cavity to remove chronic sinus disease or tumor or create access into the skullbase for extensive tumor removal. Indocyanine Green (ICG) is a dye that is injected through an intravenous site and is used to light up vasculature and margins of a tumor during surgery. This helps avoid damage to important vasculature and obtain clear margins during surgery. This study aims to further assess the utility of ICG when operating within the nasal cavity or skullbase.

DETAILED DESCRIPTION:
The investigators aim to evaluate the effectiveness and feasibility of using a fluorescent dye, Indocyanine Green (ICG), in endoscopic sinus, skullbase, sinus tumor resection, or posterior epistaxis surgery.

Adults 19 years or older, seen in the Principal Investigator and Sub investigator's offices presenting with either CRS, benign or malignant sinonasal, skull base tumors, or posterior epistaxis will be identified by the Principal Investigators and invited to participate in this prospective study. Patients will be recruited into the study in a consecutive manner. After providing consent, baseline characteristics will be collected. The investigators aim to recruit 10 patients in each study group respectively given the patients diagnosis.

Sinus tumor resection - Initially margins will be estimated with the naked eye. Then they will be compared to the margins that are fluorescing with the dye.

Skull base tumor resection - The investigators will use a part of the participant's septum for the reconstruction. The investigators will measure the time it takes for the flap to fluoresce and ensure that it is still lighting up at the end of the surgery. This means that it is still receiving a good supply and ensures longevity of the flap.

Sinus Surgery - During the participant's surgery, the investigator will come across important vessels that will be preserved. The investigator will see if the ICG is able to light up those vessels and if it does, then measure the time it takes to light up will be measured.

Posterior epistaxis - If a participant experiences a nose bleed that requires going into the operating room, the investigator will use ICG to locate the vessel that needs to be cauterized. The investigators will measure the time it takes for that vessel to light up.

The investigator will see the participants back on their day of surgery. During surgery, Indocyanine Green (ICG) will be injected through their intravenous line. The investigator will start with the smallest dose and increase to a dose that allows us to see the structures of interest such as vessels or tumor margins. The time it takes for a vessel or margins of a tumor to light up will be measured. Intra-operative data specific to each type of surgery being performed will be collected.

Dose-Escalation Protocol Intravenous injection

* 1.25mg (0.5mL)
* 2.5mg (1mL)
* 3.75mg (1.5mL)
* 5mg (2mL)
* 6.25mg (2.5mL) [at discretion of surgeon]
* 7.5mg (3mL) [at discretion of surgeon]

Intralesional injection

* 1.25mg (0.5mL)
* 2.5mg (1mL)
* 3.75mg (1.5mL)
* 5mg (2mL)
* 6.25mg (2.5mL) [at discretion of surgeon]
* 7.5mg (3mL) [at discretion of surgeon]

Descriptive statistics (count, absolute frequency, and 95% confidence interval) will be used to analyze the baseline characteristic data.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing skull base surgery with nasoseptal flap reconstruction.
* All patients undergoing endoscopic sinonasal surgery for benign and malignant tumor removal.
* All patients undergoing endoscopic sinus surgery for chronic rhinosinusitis (CRS) with or without polyposis.
* All patients undergoing surgical intervention for posterior epistaxis.

Exclusion Criteria:

* Patients less than 18 years of age
* Patients whom are currently pregnant
* Patients with allergies to sodium iodide or shellfish
* Patients with previous anaphylactic reaction to ICG

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Timing of ICG administration to fluorescence of distinct structures | Intra-operatively
  During surgery, the amount of time it takes for the area of interest to fluoresce will be recorded.
Cumulative amount of ICG administrated | Intra-operatively
  The total amount of ICG administrated to reach fluorescence of distinct structure will be recorded.
Maximum Dose of ICG administrated | Intra-operatively
  The maximum does/interval of ICG administrated to reach fluorescence of distinct structure will be recorded.
Images of surgeon estimated origin & margin, ICG estimated origin & margin | Intra-operatively
  Images of the structure of interests origins and margins will be captured. Images estimated by the surgeon and ICG will be collected.

SECONDARY OUTCOMES:
Adverse Rections to ICG | Intra-operatively
  Any adverse events to ICG that are experienced will be collected.